CLINICAL TRIAL: NCT04262258
Title: Effect of a Blueberry Enriched Diet on Skeletal Muscle Progenitor Cells
Brief Title: Effects of a Blueberry Enriched Diet on the Skeletal Muscle Regenerative Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 82422
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Skeletal Muscle Disorder
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blueberry Enriched Diet (Experimental): The blueberry intervention will consist of participants ingesting two servings of 19 g freeze dried blueberry powder (equivalent to 250 g whole blueberries) daily for six weeks. Subjects will ingest the freeze dried blueberries orally. Freeze dried blueberry powder will be mixed with 8-10 ounces of water and consumed. Subjects will be asked to rinse the cup to wash any remaining blueberries off of the cup and consume the rinse water. Subjects will be given a two week supply at baseline (week 0) and a four week supply when they return for their blood draw at week 2. Subjects will be asked to return empty packets and check-off daily records as a measure of compliance.
  Interventions: Dietary Supplement: Blueberry enriched diet

INTERVENTIONS:
Dietary Supplement: Blueberry enriched diet — The blueberry intervention will consist of participants ingesting two servings of 19 g freeze dried blueberry powder (equivalent to 250 g whole blueberries) daily for six weeks. Subjects will ingest the freeze dried blueberries orally. Freeze dried blueberry powder will be mixed with 8-10 ounces of water and consumed. Subjects will be asked to rinse the cup to wash any remaining blueberries off of the cup and consume the rinse water. Subjects will be given a two week supply at baseline (week 0) and a four week supply when they return for their blood draw at week 2. Subjects will be asked to return empty packets and check-off daily records as a measure of compliance.
  Other Names: freeze dried blueberries

SUMMARY:
One of the greatest challenges faced by older adults is maintaining physical function and strength with aging. Deterioration of skeletal muscle with aging leads to loss of mobility, decreased quality of life, and ultimately loss of independence. Skeletal muscle deterioration with aging is multifactorial, with a key factor being impaired skeletal muscle regeneration following damage. Muscle regeneration is a multistep process that requires a viable population of skeletal muscle specific progenitor cells (MPCs). MPCs reside in the skeletal muscle in a dormant state until activated by stress or injury cues. Upon activation, MPCs divide, commit to the muscle cell lineage, and fuse to form new multinucleated cells or repair damaged muscle cells. In older adults this regenerative process is impaired, which amplifies skeletal muscle deterioration. The investigators demonstrated that the ability of MPCs to divide (proliferate) is reduced, while MPC death is elevated in MPCs from healthy older adults. Further, the investigators have demonstrated that impaired nutrient metabolism, cellular inflammation, and oxidative stress are key mechanisms in this age-related disruption of MPC proliferation and overall skeletal muscle health. Therapies that improve the regenerative process and nutrient metabolism as well as attenuate oxidative stress and inflammation are necessary to improve overall skeletal muscle health of older adults. Blueberries have properties that the investigators hypothesize will improve the proliferative capacity (increase cell division and reduce cell death) of MPCs. Additionally, the investigators hypothesize that consumption of blueberries will improve skeletal muscle regeneration in the aging population via improved nutrient metabolism, attenuated cellular inflammation, and reduction of oxidative stress. The hypotheses will be tested using a dietary blueberry intervention. Serum from our human subjects [blueberry enriched diet (BED)-serum] will be collected and used to treat primary human MPCs. Ultimately, the investigators hypothesize that a blueberry enriched diet provides an ideal, natural therapy to improve MPC proliferative capacity, which is necessary to attenuate skeletal muscle deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Young 21-40 y women
* old 65-79 y women

Exclusion Criteria:

* known musculoskeletal disease (e.g., rheumatoid arthritis)
* movement disorder (e.g., Parkinson's disease) or other disorder that might affect skeletal muscle mass, function, or metabolism (e.g. diabetes, cancer)
* obese (BMI ≥ 30.0 kg/m2)
* long-term treatment with exogenous hormones or other pharmacological interventions -known to or that have the potential to influence muscle mass or function (e.g. glucocorticoids)
* antibiotic use within 6 months of intervention

Ages: 21 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in number of muscle progenitor cells on the imaging hemocytometer from baseline to 6 weeks of blueberry enriched diet | serum is obtained over the course of 6 weeks. Cell number is tracked over 12 days.
  Serum obtained from women consuming the blueberry enriched diet will be pooled. Cultured muscle progenitor cells (in vitro) from young and old women (obtained from a previous study) will be treated with serum from women consuming the blueberry enriched diet. The number of cells counted will be used as a marker of cell proliferation. Cell number will be measured using a hemocytometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Metabolic Research Unit, Ithaca, New York, United States

REFERENCES:
- [Derived] Blum JE, Gheller BJ, Hwang S, Bender E, Gheller M, Thalacker-Mercer AE. Consumption of a Blueberry-Enriched Diet by Women for 6 Weeks Alters Determinants of Human Muscle Progenitor Cell Function. J Nutr. 2020 Sep 1;150(9):2412-2418. doi: 10.1093/jn/nxaa190. PMID 32678436